CLINICAL TRIAL: NCT03404596
Title: Applying mHealth to Tobacco-related Health Disparities: Enhancing Aspects of Resiliency to Aid Cessation Efforts (Time2Quit)
Brief Title: Applying mHealth to Tobacco-related Health Disparities
Acronym: Time2Quit
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MCC-19002; R00MD010468 (NIH)
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Smoking Cessation
Keywords: cigarettes; quit smoking; nicotine; mindfulness; mHealth; mobile health
MeSH Terms: conditions — Smoking Cessation | interventions — Tobacco Use Cessation Devices; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Smoking Cessation Therapy (Experimental): Participants will receive 6 weeks of the nicotine patch therapy and brief counseling sessions. Participants will also receive mindfulness strategies for 10 days during both the pre- and post-quit periods via smartphone to aid in their cessation attempt. AutoSense will be worn to detect stress and lapse throughout the 10 day period.
  Interventions: Drug: Nicotine Patch; Behavioral: Counseling; Behavioral: Smartphone; Other: AutoSense

INTERVENTIONS:
Drug: Nicotine Patch — Nicotine patches and thorough education of the indications for the patch will be provided to all participants.
Behavioral: Counseling — Brief counseling sessions, 10-15 minutes each.
Behavioral: Smartphone — Ecological momentary assessment (EMA) assesses participants' moment-to-moment subjective experiences via self-report assessments on a smart phone. Participants will receive mindfulness strategies for 10 days pre- and post-quit via smart phone to aid in their cessation attempt. Text messages will be sent to provided study phones throughout the day. These messages will be short (1-3 minutes long) and will ask participants to do things like focus on the present moment, pay attention to their breathing, and be aware of their current thoughts.
Other: AutoSense — Participants will be asked to wear equipment throughout the day that will measure their physiology and smoking behavior. AutoSense unobtrusively and objectively collects physiological and behavioral data (i.e., negative affect (NA), self-regulatory capacity (SRC), and smoking) via wearable chest and wrist sensors.

SUMMARY:
The purpose of this study is to better understand what happens when someone attempts to quit smoking.

DETAILED DESCRIPTION:
Investigators will provide participants with nicotine patches, smoking cessation treatment that will include brief counseling sessions (10-15 minutes each), and text messages sent to their provided study phone throughout the day. These messages will be short (1-3 minutes long) and will ask participants to do things like focus on the present moment, pay attention to their breathing, and be aware of their current thoughts. Participants will be asked to wear equipment throughout the day that will measure their physiology and smoking behavior. Mobile Health (mHealth) is a general term for the use of mobile phones and other wireless technology in medical care.

The key outcome and hypothesized mechanisms (i.e., lapse and stress) will be measured objectively and automatically using AutoSense. AutoSense is a type of human sensing technology that allows investigators to detect smoking behavior and stress objectively through a chest strap and wrist bands worn by participants. Ecological momentary assessment (EMA) will assess acute precipitants such as negative affect, craving, self-efficacy, motivation, alcohol consumption, etc. Questionnaires will assess other predictors and mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Smoked a minimum of 3 cigarettes per day over the past year
* Expired carbon monoxide reading ≥ 6
* Motivated to quit within the next 30 days
* Valid home address
* Functioning telephone number
* Can speak, read, and write in English
* At least marginal health literacy

Exclusion Criteria:

* Contraindication for the nicotine patch (e.g., heart attack, angina, skin allergies) unless a doctor's note is provided
* Endorse current psychosis
* Have a pacemaker or implanted device
* Physically unable to wear equipment and provide a good reading of physiological measures
* Current use of tobacco cessation medications
* Current use of of smoking products other than cigarettes and e-cigarettes
* Involvement in a smoking program or currently trying to quit
* Pregnancy or lactation
* Another household member being enrolled in the study
* No prior experience with a smart phone
* The study staff or principal investigator (PI) have serious concerns about the participant's ability to engage in and/or complete the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Rate of Smoking Lapse | Up to 36 months
  Lapse will be measured objectively and automatically from the equipment worn by participants (AutoSense).
Rate of Stress | Up to 36 months
  Stress will be measured objectively and automatically from the equipment worn by participants (AutoSense).

CONTACTS AND LOCATIONS:
Overall Officials: Christine Vinci, Ph.D, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Vinci C, Sutton SK, Yang MJ, Jones SR, Kumar S, Wetter DW. Proximal Effects of a Just-in-Time Adaptive Intervention for Smoking Cessation With Wearable Sensors: Microrandomized Trial. JMIR Mhealth Uhealth. 2025 Mar 19;13:e55379. doi: 10.2196/55379. PMID 40106803
- [Derived] Hernandez LM, Wetter DW, Kumar S, Sutton SK, Vinci C. Smoking Cessation Using Wearable Sensors: Protocol for a Microrandomized Trial. JMIR Res Protoc. 2021 Feb 24;10(2):e22877. doi: 10.2196/22877. PMID 33625366
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/